CLINICAL TRIAL: NCT02718300
Title: A Phase 2 Study of the Safety, Tolerability, and Efficacy of INCB050465 in Combination With Ruxolitinib in Subjects With Myelofibrosis
Brief Title: A Study of INCB050465 in Combination With Ruxolitinib in Subjects With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A business decision was made to discontinue further enrollment. There were no safety concerns that contributed to this decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 50465-201; Parsaclisib (Other: Incyte Corporation)
Expanded Access: NCT03147742 (Approved for marketing)
Record Dates: First submitted 2016-03-21; First posted 2016-03-24 (Estimated); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: MPN (Myeloproliferative Neoplasms)
Keywords: Primary myelofibrosis (PMF); post-polycythemia vera myelofibrosis (PPV-MF); post-essential thrombocythemia myelofibrosis (PET-MF); myeloproliferative neoplasms (MPNs); phosphoinositide 3-kinase (PI3K) inhibitor; Janus kinase (JAK) inhibitor
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Hereditary Sensory and Autonomic Neuropathies | interventions — parsaclisib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Ruxolitinib + Parsaclisib (Experimental): Initial cohort dose of parsaclisib added to existing stable regimen of ruxolitinib, with subsequent cohort escalations based on protocol-specific criteria.
  Interventions: Drug: Parsaclisib; Drug: Ruxolitinib
- Part 2: Ruxolitinib + Parsaclisib (Experimental): Part 2 will compare 2 doses of parsaclisib .
  Interventions: Drug: Parsaclisib; Drug: Ruxolitinib
- Part 3: Ruxolitinib + Parsaclisib (Experimental): Part 3 will compare 2 different long term dosing strategies.
  Interventions: Drug: Ruxolitinib; Drug: Parsaclisib
- Part 4: Ruxolitinib + Parsaclisib (Experimental): Part 4 will compare 2 different daily dosing strategies.
  Interventions: Drug: Ruxolitinib; Drug: Parsaclisib

INTERVENTIONS:
Drug: Parsaclisib — Up to 3 oral once a day (QD) doses of parsaclisib. Doses will be taken once daily for 8 weeks, followed by once weekly dosing at the same dose level.
  Other Names: INCB050465
  Arms: Part 1: Ruxolitinib + Parsaclisib
Drug: Parsaclisib — Two recommended oral QD doses of parsaclisib. Once daily doses of parsaclisib will be taken for 8 weeks, followed by once weekly dosing at the same dose level.
  Other Names: INCB050465
  Arms: Part 2: Ruxolitinib + Parsaclisib
Drug: Ruxolitinib — The dose of ruxolitinib will be that which the subjects had been taking for at least 8 weeks before the first dose of parsaclisib.
  Other Names: Jakafi®
Drug: Parsaclisib — 20 mg oral QD dose of parsaclisib for 8 weeks. After 8 weeks patients will take either 20 mg once weekly or 5 mg once daily.
  Other Names: INCB050465
  Arms: Part 3: Ruxolitinib + Parsaclisib
Drug: Parsaclisib — 2 dose strategies will be compared:
  1. 5 mg parsaclisib beginning on Day 1 until end of treatment.
  2. 20 mg oral QD dose of parsaclisib for 8 weeks; after 8 weeks patients will take 5 mg once daily.
  Other Names: INCB050465
  Arms: Part 4: Ruxolitinib + Parsaclisib

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and efficacy of the combination of parsaclisib and ruxolitinib in subjects with myelofibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis, post-polycythemia vera myelofibrosis, or post-essential thrombocythemia myelofibrosis
* Palpable spleen of > 10 cm below the left subcostal margin on physical examination at the screening visit OR
* Palpable splenomegaly of 5 to 10 cm below left subcostal margin on physical exam AND active symptoms of MF at the screening visit as demonstrated by presence of 1 symptom score ≥ 5 or 2 symptom scores ≥ 3 using the Screening Symptom Form
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Use of experimental drug therapy for myelofibrosis, or any other standard drug (eg, danazol, hydroxyurea, etc) with the exception of ruxolitinib within 6 months of starting study (combination) therapy and/or lack of recovery from all toxicities from previous therapy (except ruxolitinib) to Grade 1 or better
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications
* Unwillingness to be transfused with blood components
* Recent history of inadequate bone marrow reserve as demonstrated by the following:

  * Platelet count < 50 × 10^9/L in the 4 weeks before screening or platelet transfusion(s) within 8 weeks before screening
  * Absolute neutrophil count levels < 0.5 × 10^9/L in the 4 weeks before screening
  * Subjects with peripheral blood blast count of > 10% at the screening or baseline hematology assessments
  * Subjects who are not willing to receive red blood cell (RBC) transfusions to treat low hemoglobin levels
* Inadequate liver function at screening as demonstrated by the following:

  * Direct bilirubin ≥ 2.0 × the upper limit of laboratory normal (ULN). (NOTE: direct bilirubin will only be determined if total bilirubin is ≥ 2.0 × ULN)
  * alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 × ULN
* Inadequate renal function at screening as demonstrated by creatinine clearance < 50 mL/min or glomerular filtration rate < 50 mL/min/1.73 m^2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, MD, Study Director — Incyte Corporation
Locations (39):
- United States (39):
  - Birmingham Hematology & Oncolgy Associates Llc, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Alta Bates Medical Center, Berkeley, California
  - City of Hope National Medical Center, Duarte, California
  - California Cancer Associates For Research and Excellence, Fresno, California
  - University of Southern California, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Pcr Oncology, Pismo Beach, California
  - California Cancer Assoc. for Research and Excellence, San Marcos, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Shands Hospital, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - McFarland Clinic, Ames, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Saint Agnes Hospital, Baltimore, Maryland
  - Cancer Center For Blood Disorders, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Rush University Medical Center, Nashville, Tennessee
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Renovatio Clinical Consultants Llc, The Woodlands, Texas
  - Va Salt Lake City Health Care System, Salt Lake City, Utah
  - Vista Oncology Inc Ps, Olympia, Washington

REFERENCES:
- [Derived] Yacoub A, Borate U, Rampal RK, Ali H, Wang ES, Gerds AT, Hobbs G, Kremyanskaya M, Winton E, O'Connell C, Goel S, Oh ST, Schiller G, McCloskey J, Palmer J, Holmes H, Hager S, Assad A, Erickson-Viitanen S, Zhou F, Daver N. Phase 2 study of add-on parsaclisib for patients with myelofibrosis and suboptimal response to ruxolitinib: final results. Blood Adv. 2024 Mar 26;8(6):1515-1528. doi: 10.1182/bloodadvances.2023011620. PMID 38290135

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted at 20 study centers in the United States. Participants who initially received weekly doses were given the option of transitioning to daily doses based on a preliminary analysis of data. All participants were analyzed according to their original treatment assignment in the Participant Flow and Baseline Characteristic module; those participants who transitioned from weekly to daily doses (n=8) were analyzed separately for specific outcome measures.
Groups:
- TG5I/M: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 milligrams (mg) twice a day (BID) to 25 mg BID for at least 8 weeks before randomization. From Day 1 to the end of Week 8, participants received oral parsaclisib 20 mg once daily (QD), followed by 5 mg QD until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
- TG5D: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 mg BID to 25 mg BID for at least 8 weeks before randomization. From Day 1, participants received oral parsaclisib 5 mg QD until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
- TG10 + TG20: Daily/Weekly Dosing: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 mg BID to 25 mg BID for at least 8 weeks before randomization. From Day 1 to the end of Week 8, participants in TG10 and TG20 received oral parsaclisib 10 mg or 20 mg QD, respectively, followed by the same dose weekly until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
Period: Overall Study
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Started (Due to early termination of the study, per the Statistical Analysis Plan, participants were combined into arms based on the dosage received regardless of what phase of the study they participated in.) | 21 | 21 | 32
Completed | 0 | 0 | 0
Not Completed | 21 | 21 | 32
Not completed — Death | 4 | 5 | 17
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Study Terminated by Sponsor | 6 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 4 | 3
Not completed — Transitioned to Rollover Study or Pursued Allogenic Transplant | 9 | 9 | 4

BASELINE CHARACTERISTICS:
Population: Due to early termination of the study, per the Statistical Analysis Plan, participants were combined into arms based on the dosage received regardless of what phase of the study they participated in.
Groups:
- Total: Total of all reporting groups
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing | Total
Number analyzed (Participants) | 21 | 21 | 32 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.33) | 69.3 (7.96) | 66.0 (8.94) | 67.5 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 17 | 39
  Male | 10 | 10 | 15 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 3 | 5
  Not Hispanic or Latino | 18 | 19 | 27 | 64
  Unknown or Not Reported | 3 | 0 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20 | 15 | 25 | 60
  Black or African American | 1 | 2 | 0 | 3
  Asian | 0 | 2 | 3 | 5
  Captured as "Other" in Database | 0 | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLTs were defined as the occurrence of any protocol-defined toxicities occurring up to and including Day 28, except those with a clear alternative explanation (e.g., disease progression, other medications) or transient (≤ 72 hours) abnormal laboratory values without associated clinically significant signs or symptoms based on investigator determination. All DLTs were assessed by the investigator using Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 criteria.
Time Frame: up to Day 28
Population: Initial Safety Population: all participants who received at least 1 dose of study drug. Treatment groups were determined according to the actual treatment the participant received regardless of assigned study drug treatment. Analysis was conducted on the Safety Population during the initial safety period. Due to early termination of the study, per the Statistical Analysis Plan, daily and weekly dosing arms were combined for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 21 | 21 | 32
Participants | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Spleen Volume Through Week 12 of the Initial Study Period as Measured by Magnetic Resonance Imaging (MRI) (or Computed Tomography [CT] Scan in Applicable Participants)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 12
Population: Initial Safety Population: all enrolled participants who received at least 1 dose of study drug. Analysis was conducted on the Safety Population during the initial safety period. Only participants with available data were analyzed. Due to early termination of the study, per the Statistical Analysis Plan, daily and weekly dosing arms were combined for efficacy analysis.
Measure: Mean (Standard Deviation); unit: centimeters cubed (cm^3)
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 20 | 17 | 29
centimeters cubed (cm^3)
  Baseline | 1779.0 (1006.75) | 2032.3 (773.45) | 2469.0 (1208.90)
  Change from Baseline at Week 12: number analyzed (Participants) | 20 | 17 | 28
  Change from Baseline at Week 12 | 383.3 (2342.09) | -276.9 (226.11) | -54.3 (312.69)

3. Primary Outcome: Percent Change From Baseline in Spleen Volume Through Week 12 as Measured by MRI (or CT Scan in Applicable Participants)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; Week 12
Population: Initial Safety Population. Analysis was conducted on the Safety Population during the initial safety period. Only participants with available data were analyzed. Due to early termination of the study, per the Statistical Analysis Plan, daily and weekly dosing arms were combined for efficacy analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 20 | 17 | 28
percent change | 9.2 (104.37) | -15.2 (10.89) | -3.1 (12.21)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.4046, Van Elteren test; stratified by ECOG Performance Status at Screening (0 or 1 versus 2)

4. Secondary Outcome: Change From Baseline in Spleen Volume Through Week 24 of the Initial Study Period as Measured by MRI (or CT Scan in Applicable Participants)
Description: Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 20 | 17 | 29
cm^3
  Baseline | 1779.0 (1006.75) | 2032.3 (773.45) | 2469.0 (1208.90)
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 14 | 20
  Change from Baseline at Week 24 | -292.6 (514.91) | -335.9 (204.19) | -37.5 (432.02)

5. Secondary Outcome: Percent Change From Baseline in Spleen Volume Through Week 24 as Measured by MRI (or CT Scan in Applicable Participants )
Description: as for outcome 3
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 15 | 14 | 20
percent change | -21.9 (24.10) | -19.0 (11.23) | -4.9 (18.81)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.7802, Van Elteren test; stratified by ECOG Performance Status at Screening (0 or 1 versus 2)

6. Secondary Outcome: Change From Baseline in the Total Symptom Score (TSS) Through Week 12 as Measured by Myelofibrosis Symptom Assessment Form (MFSAF) Version 3.0 (v3.0) Symptom Diary
Description: The MFSAF v3.0 is comprised of 19 individual symptom scores, each collected daily using an 11-point scale. The daily TSS is composed of 6 of these individual symptom scores (nights sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone/muscle pain) collected on the same day. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 6 symptom scores; scores ranged from 0 to 60, with higher scores corresponding to more severe symptoms. The Baseline TSS was defined as the average of daily total scores from the last 7 days before the first dose of INCB050465. The Week 12 TSS was the average of the daily total scores from the last 7 consecutive days before the Week 12 visit. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 16 | 16 | 28
scores on a scale
  Baseline | 17.6 (10.59) | 16.3 (12.82) | 15.2 (12.94)
  Change from Baseline at Week 12: number analyzed (Participants) | 12 | 12 | 22
  Change from Baseline at Week 12 | -6.0 (6.63) | -5.0 (11.15) | -2.1 (4.87)

7. Secondary Outcome: Percent Change From Baseline in the TSS Through Week 12 as Measured by MFSAF v3.0 Symptom Diary
Description: The MFSAF v3.0 is comprised of 19 individual symptom scores, each collected daily using an 11-point scale. The daily TSS is composed of 6 of these individual symptom scores (nights sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone/muscle pain) collected on the same day. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 6 symptom scores; scores ranged from 0 to 60, with higher scores corresponding to more severe symptoms. The Baseline TSS was defined as the average of daily total scores from the last 7 days before the first dose of INCB050465. The Week 12 TSS was the average of the daily total scores from the last 7 consecutive days before the Week 12 visit. Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 12 | 12 | 21
percent change | -37.0 (30.93) | -17.7 (57.81) | 10.1 (118.94)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.6856, Van Elteren test; stratified by ECOG Performance Status at Screening (0 or 1 versus 2)

8. Secondary Outcome: Change From Baseline in the TSS Through Week 24 as Measured by MFSAF v3.0 Symptom Diary
Description: The MFSAF v3.0 is comprised of 19 individual symptom scores, each collected daily using an 11-point scale. The daily TSS is composed of 6 of these individual symptom scores (nights sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone/muscle pain) collected on the same day. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 6 symptom scores; scores ranged from 0 to 60, with higher scores corresponding to more severe symptoms. The Baseline TSS was defined as the average of daily total scores from the last 7 days before the first dose of INCB050465. The Week 24 TSS was the average of the daily total scores from the last 7 consecutive days before the Week 24 visit. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 16 | 16 | 28
scores on a scale
  Baseline | 17.6 (10.59) | 16.3 (12.82) | 15.2 (12.94)
  Change from Baseline at Week 24: number analyzed (Participants) | 8 | 10 | 17
  Change from Baseline at Week 24 | -5.6 (8.97) | -3.9 (13.63) | -2.0 (7.15)

9. Secondary Outcome: Percent Change From Baseline in the TSS Through Week 24 as Measured by MFSAF v3.0 Symptom Diary
Description: The MFSAF v3.0 is comprised of 19 individual symptom scores, each collected daily using an 11-point scale. The daily TSS is composed of 6 of these individual symptom scores (nights sweats, itchiness, abdominal discomfort, pain under left ribs, early satiety, bone/muscle pain) collected on the same day. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 6 symptom scores; scores ranged from 0 to 60, with higher scores corresponding to more severe symptoms. The Baseline TSS was defined as the average of daily total scores from the last 7 days before the first dose of INCB050465. The Week 24 TSS was the average of the daily total scores from the last 7 consecutive days before the Week 24 visit. Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 8 | 10 | 16
percent change | -29.2 (41.08) | -16.7 (76.27) | 11.1 (80.23)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.3385, Van Elteren test; stratified by ECOG Performance Status at Screening (0 or 1 versus 2)

10. Secondary Outcome: Change From Baseline in the TSS Through Week 12 as Measured by Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF)
Description: The MPN-SAF weekly total score is defined as the sum of 10 individual symptom scores (fatigue, nights sweats, itchiness, bone pain, fever, unintentional weight loss last 6 months, early satiety, abdominal discomfort, inactivity, problems with concentration) collected at the same visit using an 11-point scale. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 10 symptom scores; scores ranged from 0 to 100, with higher scores corresponding to more severe symptoms. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 18 | 19 | 28
scores on a scale
  Baseline | 30.0 (17.88) | 27.7 (18.18) | 29.2 (19.56)
  Change from Baseline at Week 12: number analyzed (Participants) | 14 | 16 | 21
  Change from Baseline at Week 12 | -10.6 (12.63) | -12.6 (15.52) | -4.8 (9.78)

11. Secondary Outcome: Percent Change From Baseline in the TSS Through Week 12 as Measured by MPN-SAF
Description: The MPN-SAF weekly total score is defined as the sum of 10 individual symptom scores (fatigue, nights sweats, itchiness, bone pain, fever, unintentional weight loss last 6 months, early satiety, abdominal discomfort, inactivity, problems with concentration) collected at the same visit using an 11-point scale. Participants scored each symptom using a scale from 0 (absent) to 10 (worst imaginable). The TSS was calculated as a sum of all 10 symptom scores; scores ranged from 0 to 100, with higher scores corresponding to more severe symptoms. Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] / Baseline value) x 100.
Time Frame: Baseline; Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 14 | 16 | 20
percent change | -28.7 (42.48) | -38.1 (44.76) | -20.1 (40.88)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.4005, Van Elteren test; stratified by Easter Cooperative Oncology Group (ECOG) Performance Status at Screening (0 or 1 versus 2)

12. Secondary Outcome: Change From Baseline in the TSS Through Week 24 as Measured by MPN-SAF
Description: as for outcome 10
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 18 | 19 | 28
scores on a scale
  Baseline | 30.0 (17.88) | 27.7 (18.18) | 29.2 (19.56)
  Change from Baseline at Week 24: number analyzed (Participants) | 13 | 13 | 16
  Change from Baseline at Week 24 | -15.6 (9.95) | -12.6 (16.46) | -10.3 (11.88)

13. Secondary Outcome: Percent Change From Baseline in the TSS Through Week 24 as Measured by MPN-SAF
Description: as for outcome 11
Time Frame: Baseline; Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 13 | 13 | 15
percent change | -63.4 (28.14) | -44.7 (38.07) | -35.9 (40.43)
Statistical Analysis 1: Comparison: TG5I/M vs TG5D; Test type: Superiority; p = 0.3138, Van Elteren test; stratified by ECOG Performance Status at Screening (0 or 1 versus 2)

14. Secondary Outcome: Number of Participants With the Indicated Patient Global Impression of Change (PGIC) Score at Week 12, Week 24, and the End of Treatment (EOT)
Description: The PGIC questionnaire consists of a single question with 7 possible answers: "Since the start of treatment you've received in this study, your myelofibrosis symptoms are: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; 7, very much worse."
Time Frame: Baseline; up to 1494 days (EOT)
Population: Initial Safety Population. Analysis was conducted on the Safety Population during the initial safety period. Due to early termination of the study, per the Statistical Analysis Plan, daily and weekly dosing arms were combined for efficacy analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 21 | 21 | 32
Participants
  Week 12, very much improved | 1 | 1 | 1
  Week 12, much improved | 4 | 4 | 8
  Week 12, minimally improved | 5 | 6 | 5
  Week 12, no change | 6 | 6 | 6
  Week 12, minimally worse | 2 | 0 | 3
  Week 12, much worse | 0 | 0 | 1
  Week 12, very much worse | 0 | 0 | 0
  Week 12, not reported | 3 | 4 | 8
  Week 24, very much improved | 1 | 1 | 3
  Week 24, much improved | 7 | 4 | 9
  Week 24, minimally improved | 4 | 6 | 4
  Week 24, no change | 3 | 1 | 3
  Week 24, minimally worse | 0 | 1 | 0
  Week 24, much worse | 0 | 0 | 0
  Week 24, very much worse | 0 | 0 | 0
  Week 24, not reported | 6 | 8 | 13
  EOT, very much improved | 0 | 0 | 1
  EOT, much improved | 2 | 6 | 4
  EOT, minimally improved | 7 | 3 | 1
  EOT, no change | 4 | 5 | 3
  EOT, minimally worse | 2 | 1 | 2
  EOT, much worse | 1 | 1 | 2
  EOT, very much worse | 0 | 0 | 1
  EOT, not reported | 5 | 5 | 18

15. Secondary Outcome: Mean PGIC Score at Week 12, Week 24, and the EOT
Description: as for outcome 14
Time Frame: up to 1494 days (EOT)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 21 | 21 | 32
scores on a scale
  Week 12: number analyzed (Participants) | 18 | 17 | 24
  Week 12 | 3.2 (1.11) | 3.0 (0.94) | 3.2 (1.28)
  Week 24: number analyzed (Participants) | 15 | 13 | 19
  Week 24 | 2.6 (0.91) | 2.8 (1.01) | 2.4 (0.96)
  EOT: number analyzed (Participants) | 16 | 16 | 14
  EOT | 3.6 (1.09) | 3.3 (1.24) | 3.8 (1.85)

16. Secondary Outcome: Best Overall Response (Percentage of Participants With Complete Response [CR] or Partial Response [PR]) for Investigator-Reported International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) Response Assessment
Description: A participant was considered as a responder if the participant had a best overall response of CR or PR. CR: (a) bone marrow (BM): age-adjusted normocellularity (AAN); < 5% blasts; ≤ grade 1 myelofibrosis (MF); (b) peripheral blood (PD): hemoglobin (Hg) ≥ 100 grams per Liter (g/L) and < upper normal limit (UNL); neutrophils ≥ 1 × 10^9/L and < UNL; (c) platelets ≥ 100 × 10^9/L and < UNL; < 2% immature myeloid cells (IMCs); (d) clinical: resolution of disease symptoms; spleen/liver not palpable; no extramedullary hematopoiesis (EMH). PR: (a) PB: Hg ≥ 100 g/L and < UNL; neutrophils ≥ 1 × 10^9/L and < UNL; platelets ≥ 100 × 10^9/L and < UNL; < 2% IMCs; (b) clinical: resolution of disease symptoms; spleen/liver not palpable; no EMH; (c) BM: AAN; < 5% blasts; ≤ Grade 1 MF; and PB: Hg ≥ 85 g/L but < 100 g/L and < UNL; neutrophils ≥ 1 × 10^9/L and < UNL; platelets ≥ 50 × 10^9/L but < 100 × 10^9/L and < UNL; < 2% IMCs.
Time Frame: Week 12 and every 12 weeks thereafter (up to 1494 days [EOT])
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 21 | 21 | 32
percentage of participants | 0.0 | 9.5 | 9.4

17. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or requird changes in the study drug(s). TEAEs were defined as AEs that began or worsened from Baseline after the first administration of study drug.
Time Frame: up to approximately 4 years
Population: Initial Safety Population. Analysis was conducted on the Safety Population during the initial safety period. Due to early termination of the study, per the Statistical Analysis Plan, daily and weekly dosing arms were combined for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | TG5I/M | TG5D | TG10 + TG20: Daily/Weekly Dosing
Number analyzed (Participants) | 21 | 21 | 32
Participants | 20 | 20 | 31

18. Secondary Outcome: Number of Participants With Any TEAE During the Transition Period
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurred after a participant provided informed consent. Abnormal laboratory values or test results occurring after informed consent constituted AEs only if they induced clinical signs or symptoms, were considered clinically meaningful, required therapy (e.g., hematologic abnormality that required transfusion), or requird changes in the study drug(s). TEAEs were defined as AEs that began or worsened from Baseline after the first administration of study drug. Participants who had been assigned to dosing arms with weekly dosing beyond Week 8 had the opportunity to transition to all daily dosing at 5 mg if agreed upon by the participant and the Investigator.
Time Frame: up to approximately 4 years
Population: Transition Safety Population. AEs were reported in the initial randomization group (TG10, TG20) if the start of the AEs occurred before transitioning to TG5D. If the start of the AEs occurred after transitioning to TG5D, they were reported in the TG5D Transition arm.
Measure: Count of Participants; unit: Participants
Groups:
- TG5D Transition: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 mg BID to 25 mg BID for at least 8 weeks before randomization. Participants randomized to receive oral parsaclisib 10 mg or 20 mg QD from Day 1 to the end of Week 8 transitioned to oral parsaclisib 5 mg QD after Week 8. Transition participants received oral parsaclisib 5 mg QD until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
Arm/Group | TG5D Transition
Number analyzed (Participants) | 8
Participants | 8

19. Secondary Outcome: Cmax of Parsaclisib
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: Pharmacokinetic (PK) Population: all treated participants who contributed plasma PK samples. Only participants with available data were analyzed. To be able to form a meaningful statistical test with enough participants, participants across all treatment groups were combined according to the dose of parsaclisib received for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomoles per Liter (nmol/L)
Groups:
- Parsaclisib 5 mg: Participants in TG5I/M received oral parsaclisib 5 mg QD from Week 8 until discontinuation criteria were met. Participants in TG5D received oral parsaclisib 5 mg QD until discontinuation criteria were met. Participants in TG10 and TG20 who were randomized to receive oral parsaclisib 10 mg or 20 mg QD transitioned to oral parsaclisib 5 mg QD after Week 8.
- Parsaclisib 10 mg: Participants in TG10 received oral parsaclisib 10 mg QD for 8 weeks, followed by the same dose weekly until discontinuation criteria were met. Other participants were randomized to receive oral parsaclisib 10 mg QD for 8 weeks but transitioned to oral parsaclisib 5 mg QD after Week 8.
- Parsaclisib 20 mg: Participants in TG5I/M recevied oral parsaclisib 20 mg QD for 8 weeks. Participants in TG20 received oral parsaclisib 20 mg QD for 8 weeks, followed by the same dose weekly until discontinuation criteria were met. Other participants were randomized to receive oral parsaclisib 20 mg QD for 8 weeks, then received 5 mg QD from Week 8 until discontinuation criteria were met.
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
nanomoles per Liter (nmol/L)
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 350 (40.8) | 734 (29.4) | 1620 (31.6)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 381 (35.9) | 762 (29.2) | 1790 (30.5)
Statistical Analysis 1: Comparison: Parsaclisib 5 mg; Week 2; Test type: Superiority; p = 0.3577, ANOVA
Statistical Analysis 2: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 2; Test type: Superiority; Geometric Mean Ratio (GMR) = 1.048, 95% CI 2-sided [0.791 to 1.388] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 2; Test type: Superiority; GMR = 1.159, 95% CI 2-sided [0.936 to 1.435] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Parsaclisib 5 mg; Week 4; Test type: Superiority; p = 0.1709, ANOVA
Statistical Analysis 5: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 4; Test type: Superiority; GMR = 1.00, 95% CI 2-sided [0.780 to 1.281] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 4; Test type: Superiority; GMR = 1.176, 95% CI 2-sided [0.955 to 1.448] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

20. Secondary Outcome: Tmax of Parsaclisib
Description: tmax was defined as the time to the maximum concentration.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: PK Population. Only participants with available data were analyzed. To be able to form a meaningful statistical test with enough participants, participants across all treatment groups were combined according to the dose of parsaclisib received for analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
hours
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 1.0 [0.8 to 3.8] | 1.0 [1.0 to 2.0] | 1.0 [0.8 to 3.9]
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 1.0 [0.8 to 4.0] | 1.0 [0.8 to 2.0] | 1.0 [0.8 to 2.0]
Statistical Analysis 1: Comparison: Parsaclisib 5 mg; Week 2; Test type: Superiority; p = 0.6693, Kruskal-Wallis
Statistical Analysis 2: Comparison: Parsaclisib 5 mg; Week 4; Test type: Superiority; p = 0.1521, Kruskal-Wallis

21. Secondary Outcome: Cmin of Parsaclisib
Description: Cmin was defined as the minimum observed plasma concentration.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
nmol/L
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 38.3 (64.7) | 44.7 (106) | 151 (60.5)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 32.6 (112) | 69.2 (53.8) | 196 (75.3)
Statistical Analysis 1: Comparison: Parsaclisib 5 mg; Week 2; Test type: Superiority; p = 0.0809, ANOVA
Statistical Analysis 2: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 2; Test type: Superiority; GMR = 0.583, 95% CI 2-sided [0.342 to 0.994] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 2; Test type: Superiority; GMR = 0.986, 95% CI 2-sided [0.658 to 1.477] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Parsaclisib 5 mg; Week 4; Test type: Superiority; p = 0.1525, ANOVA
Statistical Analysis 5: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 4; Test type: Superiority; GMR = 1.062, 95% CI 2-sided [0.604 to 1.867] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 4; Test type: Superiority; GMR = 1.504, 95% CI 2-sided [0.937 to 2.414] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

22. Secondary Outcome: AUC0-4h of Parsaclisib
Description: AUC0-4h was defined as the area under the plasma concentration-time curve from time = 0 to 4 hours post-dose.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nmol/L
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
hours * nmol/L
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 982 (39.4) | 2000 (30.5) | 4560 (30.3)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 1080 (34.7) | 2140 (28.0) | 5070 (32.1)
Statistical Analysis 1: Comparison: Parsaclisib 5 mg; Week 2; Test type: Superiority; p = 0.2873, ANOVA
Statistical Analysis 2: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 2; Test type: Superiority; GMR = 1.016, 95% CI 2-sided [0.773 to 1.336] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 2; Test type: Superiority; GMR = 1.161, 95% CI 2-sided [0.943 to 1.429] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Parsaclisib 5 mg; Week 4; Test type: Superiority; p = 0.1601, ANOVA
Statistical Analysis 5: Comparison: Parsaclisib 5 mg vs Parsaclisib 10 mg; Week 4; Test type: Superiority; GMR = 0.992, 95% CI 2-sided [0.773 to 1.274] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Parsaclisib 5 mg vs Parsaclisib 20 mg; Week 4; Test type: Superiority; GMR = 1.177, 95% CI 2-sided [0.955 to 1.452] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

23. Secondary Outcome: AUC0-t of Parsaclisib
Description: AUC0-t was defined as the area under the plasma concentration-time curve from time =0 to the last measurable concentration at time = t.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x nmol/L
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
hours x nmol/L
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 982 (39.4) | 2000 (30.5) | 4560 (30.3)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 1080 (34.7) | 2140 (28.0) | 5070 (32.1)

24. Secondary Outcome: Clast of Parsaclisib
Description: Clast was defined as the last quantifiable concentration.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
nmol/L
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 224 (31.6) | 419 (24.0) | 949 (30.1)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 249 (28.9) | 424 (31.2) | 1060 (33.5)

25. Secondary Outcome: Tlast of Parsaclisib
Description: tlast was defined as the time of the last quantifiable concentration.
Time Frame: Week 2 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Parsaclisib 5 mg | Parsaclisib 10 mg | Parsaclisib 20 mg
Number analyzed (Participants) | 15 | 12 | 28
hours
  Week 2: number analyzed (Participants) | 15 | 9 | 28
  Week 2 | 3.89 (3.87) | 3.96 (1.58) | 3.94 (2.55)
  Week 4: number analyzed (Participants) | 13 | 12 | 28
  Week 4 | 3.87 (2.94) | 3.98 (2.27) | 3.94 (2.93)

26. Secondary Outcome: Cmax of Ruxolitinib
Description: Cmax was defined as the maximum observed plasma concentration.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: PK Population. Only participants with available data were analyzed. To be able to form a meaningful statistical test with enough participants, participants across all treatment groups were combined according to the pre-Day 1 stable dose of ruxolitinib received for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Ruxolitinib 5 mg: Throughout the study, participants received a stable dose of ruxolitinib 5 mg BID.
- Ruxolitinib 10 mg: Throughout the study, participants received a stable dose of ruxolitinib 10 mg BID.
- Ruxolitinib 15 mg: Throughout the study, participants received a stable dose of ruxolitinib 15 mg BID.
- Ruxolitinib 20 mg: Throughout the study, participants received a stable dose of ruxolitinib 20 mg BID.
- Ruxolitinib 25 mg: Throughout the study, participants received a stable dose of ruxolitinib 25 mg BID.
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
nmol/L
  Day 1 | 202 (39.5) | 491 (26.3) | 579 (31.8) | 760 (40.8) | 875 (31.3)
  Week 4 | 335 (53.9) | 471 (37.6) | 704 (34.9) | 855 (42.2) | 1050 (36.8)
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg; Day 1; Test type: Superiority; p = 0.0830, ANOVA
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Day 1; Test type: Superiority; GMR = 1.218, 95% CI 2-sided [0.846 to 1.753] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Day 1; Test type: Superiority; GMR = 0.957, 95% CI 2-sided [0.654 to 1.399] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Day 1; Test type: Superiority; GMR = 0.943, 95% CI 2-sided [0.656 to 1.354] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 5: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Day 1; Test type: Superiority; GMR = 0.867, 95% CI 2-sided [0.579 to 1.298] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Ruxolitinib 5 mg; Week 4; Test type: Superiority; p = 0.2402, ANOVA
Statistical Analysis 7: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Week 4; Test type: Superiority; GMR = 0.702, 95% CI 2-sided [0.461 to 1.069] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 8: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Week 4; Test type: Superiority; GMR = 0.700, 95% CI 2-sided [0.456 to 1.073] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 9: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Week 4; Test type: Superiority; GMR = 0.638, 95% CI 2-sided [0.428 to 0.951] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 10: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Week 4; Test type: Superiority; GMR = 0.627, 95% CI 2-sided [0.397 to 0.990] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

27. Secondary Outcome: Tmax of Ruxolitinib
Description: tmax was defined as the time to the maximum concentration.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Median (Full Range); unit: hours
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
hours
  Day 1 | 1.1 [0.9 to 2.0] | 1.0 [0.5 to 2.0] | 1.0 [0.8 to 1.0] | 1.0 [0.8 to 2.0] | 1.0 [1.0 to 1.9]
  Week 4 | 1.0 [0.9 to 1.0] | 1.0 [0.8 to 1.9] | 1.0 [0.8 to 2.0] | 1.0 [0.8 to 2.0] | 1.0 [0.7 to 1.1]
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg; Day 1; Test type: Superiority; p = 0.0756, Kruskal-Wallis
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg; Week 4; Test type: Superiority; p = 0.0866, Kruskal-Wallis

28. Secondary Outcome: Cmin of Ruxolitinib
Description: Cmin was defined as the minimum observed plasma concentration.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
nmol/L
  Day 1 | 9.23 (141) | 23.5 (122) | 28.7 (226) | 25.9 (263) | 24.2 (156)
  Week 4 | 11.1 (178) | 19.5 (269) | 40.7 (187) | 40.7 (331) | 47.3 (123)
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg; Day 1; Test type: Superiority; p = 0.4287, ANOVA
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Day 1; Test type: Superiority; GMR = 1.272, 95% CI 2-sided [0.329 to 4.914] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Day 1; Test type: Superiority; GMR = 1.036, 95% CI 2-sided [0.252 to 4.251] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Day 1; Test type: Superiority; GMR = 0.702, 95% CI 2-sided [0.180 to 2.731] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 5: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Day 1; Test type: Superiority; GMR = 0.525, 95% CI 2-sided [0.118 to 2.348] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Ruxolitinib 5 mg; Week 4; Test type: Superiority; p = 0.9788, ANOVA
Statistical Analysis 7: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Week 4; Test type: Superiority; GMR = 0.879, 95% CI 2-sided [0.198 to 3.896] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 8: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Week 4; Test type: Superiority; GMR = 1.225, 95% CI 2-sided [0.270 to 5.560] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 9: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Week 4; Test type: Superiority; GMR = 0.918, 95% CI 2-sided [0.221 to 3.821] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 10: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Week 4; Test type: Superiority; GMR = 0.853, 95% CI 2-sided [0.169 to 4.299] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

29. Secondary Outcome: AUC0-4h of Ruxolitinib
Description: AUC0-4h was defined as the area under the plasma concentration-time curve from time = 0 to 4 hours post-dose.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x nmol/L
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
hours x nmol/L
  Day 1 | 440 (39.7) | 1100 (25.5) | 1310 (35.8) | 1700 (52.4) | 1890 (23.4)
  Week 4 | 718 (67.9) | 1090 (29.5) | 1730 (38.9) | 1910 (51.0) | 2300 (34.2)
Statistical Analysis 1: Comparison: Ruxolitinib 5 mg; Day 1; Test type: Superiority; p = 0.1208, ANOVA
Statistical Analysis 2: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Day 1; Test type: Superiority; GMR = 1.251, 95% CI 2-sided [0.832 to 1.879] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 3: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Day 1; Test type: Superiority; GMR = 0.992, 95% CI 2-sided [0.649 to 1.518] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 4: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Day 1; Test type: Superiority; GMR = 0.967, 95% CI 2-sided [0.645 to 1.450] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 5: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Day 1; Test type: Superiority; GMR = 0.860, 95% CI 2-sided [0.548 to 1.350] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 6: Comparison: Ruxolitinib 5 mg; Week 4; Test type: Superiority; p = 0.3218, ANOVA
Statistical Analysis 7: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 10 mg; Week 4; Test type: Superiority; GMR = 0.761, 95% CI 2-sided [0.482 to 1.200] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 8: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 15 mg; Week 4; Test type: Superiority; GMR = 0.803, 95% CI 2-sided [0.506 to 1.277] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 9: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 20 mg; Week 4; Test type: Superiority; GMR = 0.667, 95% CI 2-sided [0.432 to 1.028] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD
Statistical Analysis 10: Comparison: Ruxolitinib 5 mg vs Ruxolitinib 25 mg; Week 4; Test type: Superiority; GMR = 0.640, 95% CI 2-sided [0.390 to 1.051] — ANOVA was performed on dose-normalized PK parameters per dose level. The reference group was 5 mg QD

30. Secondary Outcome: AUC0-t of Ruxolitinib
Description: as for outcome 23
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x nmol/L
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
hours x nmol/L
  Day 1 | 440 (39.7) | 1100 (25.5) | 1310 (35.8) | 1700 (52.4) | 1890 (23.4)
  Week 4 | 718 (67.9) | 1090 (29.5) | 1730 (38.9) | 1910 (51.0) | 2300 (34.2)

31. Secondary Outcome: Clast of Ruxolitinib
Description: Clast was defined as the last quantifiable concentration.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
nmol/L
  Day 1 | 53.0 (60.4) | 145 (38.2) | 213 (64.1) | 233 (109) | 235 (38.8)
  Week 4 | 87.1 (111) | 156 (36.4) | 285 (58.7) | 270 (87.3) | 294 (48.3)

32. Secondary Outcome: Tlast of Ruxolitinib
Description: tlast was defined as the time of the last quantifiable concentration.
Time Frame: Day 1 and Week 4: predose and 1, 2, and 4 hours post-dose
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Ruxolitinib 5 mg | Ruxolitinib 10 mg | Ruxolitinib 15 mg | Ruxolitinib 20 mg | Ruxolitinib 25 mg
Number analyzed (Participants) | 4 | 18 | 12 | 19 | 8
hours
  Day 1 | 3.97 (2.72) | 3.92 (4.04) | 3.89 (4.63) | 3.99 (1.27) | 3.99 (1.20)
  Week 4 | 3.94 (2.06) | 3.92 (1.87) | 3.95 (3.57) | 3.93 (2.66) | 3.89 (3.68)

ADVERSE EVENTS:
Time Frame: up to approximately 1529 days
Description: An AE was reported in the initial randomization group (TG10, TG20) if it started before transition to TG5D. An AE was reported in the TG5D Transition arm if it started after transition to TG5D. Due to early termination of the study, per the Statistical Analysis Plan, the 4 dosage groups (TG10: Daily/Weekly Dosing; TG20: Daily/Weekly Dosing; TG5I/M; TG5D), as well as the participants who transitioned from daily/weekly to all-daily dosing (TG5D Transition), were compared separately for safety.
Groups:
- TG10: Daily/Weekly Dosing: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 mg BID to 25 mg BID for at least 8 weeks before randomization. From Day 1 to the end of Week 8, participants received oral parsaclisib 10 milligrams (mg) once daily (QD), followed by the same dose weekly until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
- TG20: Daily/Weekly Dosing: Participants received at least 6 months of prior ruxolitinib therapy, including ruxolitinib administration at a stable dose of 5 mg BID to 25 mg BID for at least 8 weeks before randomization. From Day 1 to the end of Week 8, participants received oral parsaclisib 20 mg QD, followed by the same dose weekly until discontinuation criteria were met, in combination with the pre-Day 1 stable dose of ruxolitinib (5 to 25 mg BID).
- Total: Initially Randomized Participants: Total
Arm/Group | TG10: Daily/Weekly Dosing | TG20: Daily/Weekly Dosing | TG5I/M | TG5D | Total: Initially Randomized Participants | TG5D Transition
All-Cause Mortality (participants affected / at risk) | 6/14 | 11/18 | 4/21 | 5/21 | 26/74 | 3/8
Serious Adverse Events (participants affected / at risk) | 2/14 | 11/18 | 7/21 | 6/21 | 26/74 | 3/8
Other Adverse Events (participants affected / at risk) | 13/14 | 18/18 | 20/21 | 20/21 | 71/74 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG10: Daily/Weekly Dosing (N=14) | TG20: Daily/Weekly Dosing (N=18) | TG5I/M (N=21) | TG5D (N=21) | Total: Initially Randomized Participants (N=74) | TG5D Transition (N=8)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 6 (6) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tobacco withdrawal symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG10: Daily/Weekly Dosing (N=14) | TG20: Daily/Weekly Dosing (N=18) | TG5I/M (N=21) | TG5D (N=21) | Total: Initially Randomized Participants (N=74) | TG5D Transition (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 6 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 3 (4) | 4 (4) | 3 (3) | 13 (15) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 7 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (5) | 4 (4) | 3 (5) | 13 (16) | 2 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 3 (3) | 2 (2) | 8 (9) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 0 (0)
Asthenia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 3 (3) | 1 (1) | 9 (10) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 3 (4) | 2 (2) | 2 (3) | 8 (10) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (3) | 5 (5) | 11 (14) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 6 (6) | 0 (0) | 0 (0) | 8 (8) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (9) | 4 (4) | 2 (3) | 13 (17) | 0 (0)
Cytomegalovirus viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 1 (2) | 1 (1) | 5 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 3 (5) | 3 (3) | 4 (4) | 15 (17) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4) | 4 (5) | 12 (13) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 3 (3) | 4 (5) | 12 (13) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Early satiety (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 2 (2) | 1 (1) | 9 (10) | 0 (0)
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 2 (2) | 3 (8) | 10 (16) | 3 (3)
Fatigue (General disorders) | 2 (2) | 7 (7) | 4 (4) | 1 (1) | 14 (14) | 0 (0)
Feeling abnormal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 7 (8) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 5 (6) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 5 (6) | 1 (1)
Hyperplastic cholecystopathy (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5) | 2 (2) | 4 (4) | 10 (13) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 8 (8) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Morton's neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (5) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 6 (7) | 2 (2) | 5 (5) | 16 (18) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral blood blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 6 (7) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 8 (8) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 5 (11) | 2 (8) | 3 (16) | 13 (39) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7) | 3 (3) | 2 (2) | 10 (13) | 2 (2)
Pyrexia (General disorders) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 6 (8) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 8 (8) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 5 (5) | 6 (12) | 6 (7) | 20 (27) | 2 (4)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 3 (4) | 8 (9) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 5 (7) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2018-10-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02718300/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT02718300/SAP_001.pdf